CLINICAL TRIAL: NCT01620138
Title: Somatostatin and Dopamine Receptors Expression in Non-functioning Pituitary Adenomas and Resistant Prolactinomas: Correlation With in Vitro and in Vivo Responsiveness to Somatostatin Analogs and Dopamine Agonist
Brief Title: Response to Cabergoline and Pasireotide in Non-functioning Pituitary Adenomas and Resistant Prolactinomas
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Universidade Federal do Rio de Janeiro (Other)
Responsible Party: Principal Investigator, Monica Gadelha, Principal Investigator, Universidade Federal do Rio de Janeiro
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSOM230BBR01T
Record Dates: First submitted 2011-09-18; First posted 2012-06-15 (Estimated); Results first posted 2016-06-16 (Estimated); Last update posted 2016-08-22 (Estimated); Status verified 2016-07

CONDITIONS: Non-functioning Pituitary Adenomas; Prolactinomas
Keywords: Non-functioning pituitary adenomas; Prolactinomas; Cabergoline; Pasireotide; somatostatin receptors; Dopamine receptors
MeSH Terms: conditions — Prolactinoma | interventions — pasireotide; Cabergoline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pasireotide (Active Comparator): For non-cured patients with prolactinomas resistant to cabergoline, MRI will be performed immediately before and six months after the onset of pasireotide treatment. The anti-secretory effect will be evaluated by prolactin dosage every month.
  For patients harboring a NFPA, treatment will be started at least 3 months after neurosurgery, when a pituitary MRI clearly shows the presence of a residual tumor without any possible misinterpretation of postsurgical changes. In this case, the drug efficacy will be evaluated clinically by visual field and by MRI six months after pasireotide treatment.
  Interventions: Drug: Pasireotide
- cabergoline (Active Comparator): In patients with non-functioning pituitary adenoma, treatment will be started at least 3 months after neurosurgery, when a pituitary MRI clearly shows the presence of a residual tumor without any possible misinterpretation of postsurgical changes. The drug response will be evaluated clinically by visual field and by Magnetic resonance imaging (MRI) before medical treatment and after six months of cabergoline treatment at maximum dose.
  Interventions: Drug: cabergoline

INTERVENTIONS:
Drug: Pasireotide — The patients with NFPA will be randomized into two groups: (A) the first one will be treated with pasireotide at the dosage of 900 µg s.c. twice a day for 6 months; (B) the second one, with cabergoline 3 mg/week for six months.
  The patients with resistant prolactinomas will be treated with pasireotide at the dosage of 600 µg s.c. twice a day. After four weeks of treatment, the patients who normalize serum prolactin level will be maintained at the same dosage, the others who do not achieve normal prolactin level will have their dosage raised to 900 µg s.c. twice a day for six months.
  Other Names: Signifor
  Arms: Pasireotide
Drug: cabergoline — The patients with NFPA will be randomized into two groups: (A) the first one will be treated with pasireotide at 900 µg s.c. twice a day for 6 months; (B) the second one, with cabergoline 3 mg/week for 6 months.
  The patients with resistant prolactinomas will be treated with pasireotide at 600 µg s.c. twice a day. After four weeks of treatment, the patients who normalize serum prolactin level will be maintained at the same dosage, the others who do not achieve normal prolactin level will have their dosage raised to 900 µg s.c. twice a day for six months.
  Other Names: Dostinex
  Arms: cabergoline

SUMMARY:
There are no available medical treatment options for patients with non-functioning pituitary adenomas (NFPA) or with resistant prolactinomas to dopamine agonists (DA) who are not cured by surgery. The study of the receptors by quantitative messenger ribonucleic acid (mRNA) expression levels and immunohistochemistry analysis might end with a better understanding of these tumors. Besides that, it will be assessed the in vitro and in vivo responses to pasireotide (for NFPA and prolactinomas) and cabergoline (for NFPA). These responses will be compared with the receptor expressions which may be a tool as a predicting element of the response to these compounds.

DETAILED DESCRIPTION:
The goals of this study are: to verify whether cabergoline and pasireotide are effective in NFPA to control tumor re-growth as adjuvant therapy after neurosurgery and whether pasireotide is capable of normalizing the prolactin levels in patients with prolactinomas resistant to cabergoline; to assess the mRNA levels of dopamine receptor type 2 (DR2) and SSTR1-5 and their protein expression; to evaluate the in vitro hormonal response to cabergoline, octreotide and pasireotide; and to determine whether the mRNA DR2/SSTR1-5 and/or protein expression and/or in vitro hormonal response to cabergoline, octreotide and pasireotide correlates with the in vivo response to the former and to the last one. With this data the investigators intend to establish if the mRNA analysis and/or protein expression in NFPA and resistant prolactinomas might be predictive or foretelling factors concerning drug treatment in patients with this kind of pituitary tumors and also evaluate if there is any response in vitro or in vivo to the treatment with pasireotide in NFPA and resistant prolactinomas and with cabergoline in NFPA.

ELIGIBILITY:
Inclusion Criteria

* Male or female patients aged 18 years or greater
* Patients with confirmed diagnosis of NFPA evidenced by: magnetic resonance imaging (MRI) confirmation of pituitary adenoma and No pituitary tumoral hormone hypersecretion
* Patients with no previous medical treatment
* Patients who had been submitted to surgery but not cured. Lack of cure is defined as presence of remnant tumor on MRI at least three months after surgery (without any possible misinterpretation of postsurgical changes)
* Patients with confirmed diagnosis of resistant prolactinoma by lack of prolactin normalization with a tolerated cabergoline dosage during 12 weeks
* Patients who had been submitted to surgery due to resistance to cabergoline and not cured. Lack of cure is defined as lack of serum prolactin normalization or complete removal of tumor load
* Patients who signed the informed consent

Exclusion Criteria

* Previous pituitary radiotherapy
* High risk for transsphenoidal surgery
* Patients with symptomatic cholelithiasis
* Diabetic patients on antidiabetic medications those fasting blood glucose is poorly controlled as evidenced by HbA1C > 8%
* Patients with abnormal coagulation (prothrombin time (PT) or partial thromboplastin time (PTT) elevated by 30% above normal limits);
* Patients receiving anticoagulants that affect PT or PTT
* Patients who have congestive heart failure (NYHA Class III or IV), unstable angina, sustained ventricular tachycardia, clinically significant bradycardia, advanced heart block, history of acute MI less than one year prior to study entry or clinically significant impairment in cardiovascular function
* Patients with risk factors for torsade de pointes, i.e. patients with a baseline corrected QT interval (QTc) > 480 ms, hypokalemia, family history of long QT syndrome, and concomitant medications known to prolong QT interval
* Patients with liver disease such as cirrhosis, chronic active hepatitis, or chronic persistent hepatitis, or patients with (alanine aminotransferase) ALT/ (aspartate aminotransferase) AST more than 2 X upper limit of normal (ULN), serum creatinine > 2.0 X ULN, serum bilirubin > 2.0 X ULN, serum albumin < 0.67 X lower limit of normal (LLN)
* Patients with white blood cell (WBC) < 3 X 109/L; Hgb < LLN; Platelet count (PLT) < 100 X 109/L
* Patients who have any current or prior medical condition that can interfere with the conduct of the study or the evaluation of its results in the opinion of the investigator
* Female patients who are pregnant or lactating, or are of childbearing potential and not practicing a medically acceptable method for birth control. Female patients must use barrier contraception with condoms. If oral contraception is used, the patient must have been practicing this method for at least two months prior to enrollment and must agree to continue the oral contraceptive throughout the course of the study and for one month after the last dose of study drug. Male patients who are sexually active are required to use condoms during the study and for 1 month afterwards
* Patients who have a history of alcohol or drug abuse in the 6 month period prior to receiving pasireotide

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2010-03; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mônica R. Gadelha, PhD, Principal Investigator — Endocrinology Section - Hospital Universitário Clementino Fraga Filho/Federal University of Rio de Janeiro
Locations (1):
- Endocrinology Section - Hospital Universitário Clementino Fraga Filho/Federal University of Rio de Janeiro, Rio de Janeiro, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Pasireotide: Non-cured patients with resistant prolactinomas, MRI will be performed immediately before and six months after the onset of pasireotide. The efficacy will be evaluated by prolactin dosage every month.
  Patients with a nonfunctioning pituitary adenoma (NFPA), treatment will be started at least 3 months after neurosurgery. The efficacy will be evaluated by MRI 6 months after pasireotide.
  Pasireotide: The patients with NFPA will be randomized into two groups: (A) the first one will be treated with pasireotide at the dosage of 900 µg s.c. twice a day for 6 months; (B) the second one, with cabergoline 3 mg/week for 6 months.
  The patients with resistant prolactinomas will be treated with pasireotide at the dosage of 600 µg s.c. twice a day. After 4 weeks of treatment, the patients who normalize serum prolactin level will be maintained at the same dosage, the others who do not achieve normal prolactin level will have their dosage raised to 900 µg s.c. twice a day for 6 months.
- Cabergoline: In patients with non-functioning pituitary adenoma, treatment will be started at least 3 months after neurosurgery. The drug response will be evaluated clinically by visual field and by Magnetic resonance imaging (MRI) before medical treatment and after six months of cabergoline treatment at maximum dose.
  cabergoline: The patients with NFPA will be randomized into two groups: (A) the first one will be treated with pasireotide at 900 µg s.c. twice a day for 6 months; (B) the second one, with cabergoline 3 mg/week for 6 months.
  The patients with resistant prolactinomas will be treated with pasireotide at 600 µg s.c. twice a day. After four weeks of treatment, the patients who normalize serum prolactin level will be maintained at the same dosage, the others who do not achieve normal prolactin level will have their dosage raised to 900 µg s.c. twice a day for six months.
Period: Overall Study
Arm/Group | Pasireotide | Cabergoline
Started | 12 | 9
Completed | 6 | 9
Not Completed | 6 | 0
Not completed — Withdrawal by Subject | 3 | 0
Not completed — Lack of Efficacy | 1 | 0
Not completed — Adverse Event | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Pasireotide: For non-cured patients with resistant prolactinomas , MRI will be performed before and six months after the onset of pasireotide. The efficacy will be evaluated by prolactin dosage every month.
  For patients harboring a NFPA, treatment will be started at least 3 months after neurosurgery. In this case, the drug efficacy will be evaluated clinically by MRI six months after pasireotide.
  Pasireotide: The patients with NFPA will be randomized into two groups: (A) the first one will be treated with pasireotide at the dosage of 900 µg s.c. twice a day for 6 months; (B) the second one, with cabergoline 3 mg/week for six months.
  The patients with resistant prolactinomas will be treated with pasireotide at the dosage of 600 µg s.c. twice a day. After four weeks of treatment, the patients who normalize serum prolactin level will be maintained at the same dosage, the others who do not achieve normal prolactin level will have their dosage raised to 900 µg s.c. twice a day for six months.
- Total: Total of all reporting groups
Arm/Group | Pasireotide | Cabergoline | Total
Number analyzed (Participants) | 12 | 9 | 21
Age, Continuous [Median (Full Range); unit: years] | 33 [24 to 63] | 54 [36 to 65] | 54 [24 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 5 | 13
  Male | 4 | 4 | 8
Region of Enrollment [Number; unit: participants]
  Brazil | 12 | 9 | 21

OUTCOME MEASURES:

1. Primary Outcome: Tumor Volume Changes for NFPA and Prolactin Level Changes for Prolactinoma
Description: Magnetic resonance imaging (MRI) of the sella and prolactin will be performed before (baseline) and after 6 months of treatment with cabergoline or pasireotide. Disease progression will be defined as tumor growth > 25%, stable disease as changes < 25% and significant tumor shrinkage as > 25% in tumor volume compared to baseline MRI (baseline to six months).
Time Frame: Baseline to six months
Measure: Median (Full Range); unit: cmˆ3
Groups:
- Pasireotide: For non-cured patients with resistant prolactinomas, MRI will be performed immediately before and six months after the onset of pasireotide. The efficacy will be evaluated by prolactin dosage every month.
  For patients harboring a NFPA, treatment will be started at least 3 months after neurosurgery. In this case, the drug efficacy will be evaluated by MRI six months after pasireotide.
  Pasireotide: The patients with NFPA will be randomized into two groups: (A) the first one will be treated with pasireotide at the dosage of 900 µg s.c. twice a day for 6 months; (B) the second one, with cabergoline 3 mg/week for six months.
  The patients with resistant prolactinomas will be treated with pasireotide at the dosage of 600 µg s.c. twice a day. After four weeks of treatment, the patients who normalize serum prolactin level will be maintained at the same dosage, the others who do not achieve normal prolactin level will have their dosage raised to 900 µg s.c. twice a day for six months.
Arm/Group | Pasireotide | Cabergoline
Number analyzed (Participants) | 6 | 9
cmˆ3 | 3.8 [3.46 to 4.58] | 29.35 [2.55 to 51.93]
Statistical Analysis 1: Comparison: Pasireotide vs Cabergoline; Test type: Superiority or Other; p < 0.05, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Groups:
- Pasireotide: For non-cured patients with resistant prolactinomas , MRI will be performed immediately before and six months after the onset of pasireotide . The efficacy will be evaluated by prolactin dosage every month.
  For patients harboring a NFPA, treatment will be started at least 3 months after neurosurgery. In this case, the drug efficacy will be evaluated by MRI six months after pasireotide.
  Pasireotide: The patients with NFPA will be randomized into two groups: (A) the first one will be treated with pasireotide at the dosage of 900 µg s.c. twice a day for 6 months; (B) the second one, with cabergoline 3 mg/week for six months.
  The patients with resistant prolactinomas will be treated with pasireotide at the dosage of 600 µg s.c. twice a day. After four weeks of treatment, the patients who normalize serum prolactin level will be maintained at the same dosage, the others who do not achieve normal prolactin level will have their dosage raised to 900 µg s.c. twice a day for six months.
Arm/Group | Pasireotide | Cabergoline
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/9
Other Adverse Events (participants affected / at risk) | 2/12 | 0/9
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pasireotide (N=12) | Cabergoline (N=9)
Hyperglycemia (Endocrine disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No